CLINICAL TRIAL: NCT07351331
Title: The Effectiveness of Intratissue Percutaneous Electrolysis in the Shortening of the Flexor Hallucis Brevis Caused by Myofascial Pain Syndrome. A Pre-post Study.
Brief Title: Intratissue Electrolysis (EPI) is Effective in Deactivating Myofascial Trigger Points (MTrPs). (EPIEMG)
Acronym: EPIEMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPIEMG
Record Dates: First submitted 2025-11-17; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Pain Syndrome (MPS)
Keywords: Percutaneous electrolysis; Dry needling; Myofascial pain syndrome; Flexor hallucis brevis; Electromyography; Pressure platform
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Percutaneous Intratisular Electrolysis (IPE) (Experimental): To perform the intervention correctly, whether for DN or IPE, the patient is positioned in a prone position. followed by disinfection with an antiseptic applied to the region to be addressed, with the therapist always wearing gloves as protection. Once the respective treatment is completed, pressure is applied to the needle entry point for 30 seconds. The IPE intervention is performed with the Physio Invasiva® device (Enraf Nonius Ibérica S.A., Madrid, Spain), following the same approach as in the DN, with gloves worn and the region disinfected beforehand. The tense band is located to introduce the needle into the nodule, attempting to elicit a LTR produced by an MTP (20,34,37,38) , Galvanic current is then applied, with 3 pulses of 5 seconds each at an intensity of 1.5 milliamperes (mA) and current interruption between each pulse (34) , differing from other studies that apply 3 mA or more (37,38) .
  Interventions: Other: Intratissue Percutaneous Electroly
- dry needling (DN) (Experimental): To perform the intervention correctly, whether for DN or IPE, the patient is positioned in a prone position. followed by disinfection with an antiseptic applied to the region to be addressed, with the therapist always wearing gloves as protection. Once the respective treatment is completed, pressure is applied to the needle entry point for 30 seconds. The intervention with DN is performed using the "quick entries and exits technique of Hong" (35) , with gloves and alcohol disinfectant applied to the region to be treated, in this case, the internal part of the plantar foot (FHB) (33) . Next, the taud band of the FHB muscle is located, and a palpable nodule that is painful to mechanical stimulation is identified in the taud band. The needle is then inserted into the nodule to perform the "quick entry and exit technique" (34) , with 4 entries and exits performed on the FHB, aiming to provoke local twich responses (LTR)
  Interventions: Other: dry needling

INTERVENTIONS:
Other: Intratissue Percutaneous Electroly — Three interventions were performed, the first in the initial week, after pressure and sEMG measurements, the second in week 4, and the third in week 12.
  Arms: Group Percutaneous Intratisular Electrolysis (IPE)
Other: dry needling — Three interventions were performed, the first in the initial week, after pressure and sEMG measurements, the second in week 4, and the third in week 12.
  Arms: dry needling (DN)

SUMMARY:
Invasive physiotherapy techniques, such as Intratissue Percutaneous Electroly-sis (IPE), have numerous beneficial effects depending on the pathology being treated, in-cluding the deactivation of myofascial trigger points (MTP) caused by myofascial pain syndrome (MPS).

The objectives are (1) evaluate the effectiveness of low intesity IPE treatment com-pared to DN on the shortening of FHB in patients with MPS, in 4 and 12 weeks evaluation, (2) assess the distribution of plantar pressures after the interventions and (3) evaluate the modification of FHB activation following the interventions.

DETAILED DESCRIPTION:
Patients are divided into two intervention groups (IPE; n=18) and (DN; n=22). Before the intervention, variables of mean and maximum pressure are measured in all patients using a pressure platform, and neuromuscular activity is assessed through surface electromy-ography (sEMG). These measures are repeated at 4- and 12-weeks post-intervention. The results show efficacy in both techniques, with significant differences at both 4 weeks and 12 weeks in favor of the IPE group, both in plantar pressure distribution and muscular activity.

The first measurement (week of November 25, 2024) is considered the baseline measurement since the subjects had not been previously intervened. Therefore, the measurement is first performed using the pressure platform and sEMG, followed by the intervention of DN or IPE based on the group to which the subjects were previously as-signed.

At week 4 from the first measurement (week of December 23, 2024), the second data collection is conducted, using the same procedure as in the first measurement.

At week 12 from the initial measurement (week of February 17, 2025), the third data collection takes place using the same procedure as the previous two, with the difference that in this final measurement there will be no intervention of DN or IPE.

ELIGIBILITY:
Inclusion Criteria:

* subjects with ages between 18 and 65 years,
* hypersensitive spot within a taut band in FHB muscle.
* pain upon stimulation of the MTP.
* painful limit to the full range of motion

Exclusion Criteria:

* subjets who had bilateral LTP present.
* who have had a lower limb injury or surgery within the last 6 months.
* subjectss with active pathologies at the time of measurement in the lower limb.
* subjectss with cognitive impairment.
* subjectss with belonephobia or contraindications for the use of needles (oral anticoagulant therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
mean pressures (MP) | It was measured at the start of the protocol in week 1, in week 4 and in week 12.
  it is the average value of the pressure measured on a pressure platform, representing the general distribution of force per unit area across a surface (g/cm²)
maximum pressures (PMáx) | It was measured at the start of the protocol in week 1, in week 4 and in week 12.
  it is the highest pressure value recorded on the pressure platform, indicating the point of greatest concentration of force per unit area on the evaluated surface.(g/cm²)
maximal voluntary contraction (MVC) | It was measured at the start of the protocol in week 1, in week 4 and in week 12.
  The muscular activation is analyzed during 3 sets of 5 seconds of isometric contraction, against the resistance of the examiner's hand
dynamic muscular activation of the FHB | It was measured at the start of the protocol in week 1, in week 4 and in week 12.
  The subject's position is a protocol that has been previously explained to ensure correct measurement. The subject must walk for 20 seconds

CONTACTS AND LOCATIONS:
Overall Officials: María de Pedro Benito, PhD, Study Director — Associate Professor
Locations (1):
- Universidad Camilo José Cela, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martinez-Jimenez EM, Losa-Iglesias ME, Antolin-Gil MS, Lopez-Lopez D, Romero-Morales C, Benito-de-Pedro M, Calvo-Lobo C, Becerro-de-Bengoa-Vallejo R. Flexor Digitorum Brevis Muscle Dry Needling Changes Surface and Plantar Pressures: A Pre-Post Study. Life (Basel). 2021 Jan 13;11(1):48. doi: 10.3390/life11010048. PMID 33451013
- [Result] Rodriguez-Huguet M, Gongora-Rodriguez J, Rodriguez-Huguet P, Ibanez-Vera AJ, Rodriguez-Almagro D, Martin-Valero R, Diaz-Fernandez A, Lomas-Vega R. Effectiveness of Percutaneous Electrolysis in Supraspinatus Tendinopathy: A Single-Blinded Randomized Controlled Trial. J Clin Med. 2020 Jun 12;9(6):1837. doi: 10.3390/jcm9061837. PMID 32545583
- [Result] Martinez-Jimenez EM, Losa-Iglesias ME, Mazoteras-Pardo V, Lopez-Lopez D, Pereiro-Buceta H, Calvo-Lobo C, Rodriguez-Sanz D, Becerro-de-Bengoa-Vallejo R, Navarro-Flores E. Dry needling of the flexor digitorum brevis muscle reduces postural control in standing: A pre-post stabilometric study. J Anat. 2023 Sep;243(3):545-554. doi: 10.1111/joa.13862. Epub 2023 Mar 16. PMID 36924312
- [Result] Benito-de-Pedro AI, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Rodriguez-Sanz D, Calvo-Lobo C, Benito-de-Pedro M. Efficacy of Deep Dry Needling versus Percutaneous Electrolysis in Ultrasound-Guided Treatment of Active Myofascial Trigger Points of the Levator Scapulae in Short-Term: A Randomized Controlled Trial. Life (Basel). 2023 Apr 3;13(4):939. doi: 10.3390/life13040939. PMID 37109468
- [Result] Lopez-Martos R, Gonzalez-Perez LM, Ruiz-Canela-Mendez P, Urresti-Lopez FJ, Gutierrez-Perez JL, Infante-Cossio P. Randomized, double-blind study comparing percutaneous electrolysis and dry needling for the management of temporomandibular myofascial pain. Med Oral Patol Oral Cir Bucal. 2018 Jul 1;23(4):e454-e462. doi: 10.4317/medoral.22488. PMID 29924769
- [Result] Galasso A, Urits I, An D, Nguyen D, Borchart M, Yazdi C, Manchikanti L, Kaye RJ, Kaye AD, Mancuso KF, Viswanath O. A Comprehensive Review of the Treatment and Management of Myofascial Pain Syndrome. Curr Pain Headache Rep. 2020 Jun 27;24(8):43. doi: 10.1007/s11916-020-00877-5. PMID 32594264